CLINICAL TRIAL: NCT00417625
Title: Validation of Cardiac MR Perfusion With Cardiac Catheterization Physiological Assessment
Brief Title: Validation of MRI Measurement of Cardiac Blood Flow
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070056; 07-H-0056
Record Dates: First submitted 2006-12-30; First posted 2007-01-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-07-19

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Perfusion; MRI; Fractional Flow Reserve; Coronary Flow Reserve; Collateral Artery Perfusion; Cardiovascular Disease; Coronary Artery Disease; CAD
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will test the accuracy of magnetic resonance imaging (MRI) in measuring cardiac perfusion (blood flow). MRI of the heart can measure blood flow to heart muscle, but collateral coronary arteries (vessels that supply blood to the heart muscle) may reduce the accuracy of the measurements. This study will perform special measurements of coronary artery flow and pressure in patients undergoing heart catheterization and catheter-based treatment (angioplasty and stenting) in order to compare for accuracy with cardiac MRI.

Patients 21 years of age and older with coronary artery blockage may be eligible for this study. All participants undergo cardiac MRI, to produce images of the heart, as well as special invasive blood flow testing during heart catheterization, angioplasty, and stenting.

During MRI, the subject lies on a table that can slide in and out of the scanner (a narrow cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The procedure lasts about 45 to 90 minutes. Since the heart moves during breathing, subjects are asked to hold their breath intermittently for about 5-20 seconds. A medicine called dipyridamole is injected through a vein in the subject's arm to increase blood flow to the coronary arteries and help detect blockages. Pictures are taken of the heart before, during, and after the dipyridamole injection. Another medicine called gadolinium is also given through a vein. This medicine brightens the images to measure blood flow.

During a separate catheterization, angioplasty, and stenting procedure, subjects undergo additional invasive tests. The additional tests use a special guidewire to measure coronary artery pressure and blood flow, as well as a special ultrasound to look inside the artery.

Patients have a repeat MRI about 2 months after the catheterization.

DETAILED DESCRIPTION:
Cardiac magnetic resonance imaging (MRI) can measure perfusion (blood flow) to heart muscle. Collateral coronary arteries (natural bypasses to the heart) may reduce the accuracy of perfusion measured by cardiac MRI.

We are testing the accuracy of these measurements in subjects undergoing medically necessary cardiac catheterization and catheter-based treatment (angioplasty and stenting). We will perform special invasive measurements of coronary artery flow and pressure during catheterization in order to compare with cardiac MRI.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with known or suspected cardiovascular disease
* Age above age 21 (coronary artery disease is rare in subjects less than age 21)
* Undergoing medically necessary coronary arteriography
* Written informed consent
* The subject must allow access to the use of previous medical information from NIH or any institution in order to participate in the research study.

EXCLUSION CRITERIA:

Medical Exclusion Criteria:

* Pregnant women (when uncertain, subjects will undergo urine or blood testing) or lactating women
* Decompensated congestive heart failure (unable to lie flat during MRI or catheterization)
* Impaired renal excretory function (calculated Glomerular Filtration Rate less than 30mL/min/1.73m(2)) unless on dialysis.

MRI Exclusion Criteria (for MRI scan only):

* Cardiac pacemaker or implantable defibrillator
* Cerebral aneurysm clip
* Neural stimulator (e.g. TENS-Unit)
* Any type of ear implant
* Ocular foreign body (e.g. metal shavings)
* Any implanted device (e.g. insulin pump, drug infusion device)
* Metal shrapnel or bullet.

Unable to tolerate dipyridamole:

-Reactive airways disease (significant asthma or chronic obstructive pulmonary disease and unable to tolerate a beta adrenergic antagonist).

Post-Hoc Catheterization Exclusion Criteria (determined during coronary arteriography):

* Excessive tortuosity or any angiographic features that, in the opinion of catheterization operator, would make invasive physiology assessments unsafe or unsuitable
* Ongoing myocardial ischemia or other exigency that would make further study participation hazardous
* Normal epicardial coronary arteries and normal perfusion cardiac MRI

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-12-29; Study Completion 2010-07-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Muehling OM, Jerosch-Herold M, Panse P, Zenovich A, Wilson BV, Wilson RF, Wilke N. Regional heterogeneity of myocardial perfusion in healthy human myocardium: assessment with magnetic resonance perfusion imaging. J Cardiovasc Magn Reson. 2004;6(2):499-507. doi: 10.1081/jcmr-120030570. PMID 15137334
- [Background] Jerosch-Herold M, Swingen C, Seethamraju RT. Myocardial blood flow quantification with MRI by model-independent deconvolution. Med Phys. 2002 May;29(5):886-97. doi: 10.1118/1.1473135. PMID 12033585
- [Background] Muhling OM, Dickson ME, Zenovich A, Huang Y, Wilson BV, Wilson RF, Anand IS, Seethamraju RT, Jerosch-Herold M, Wilke NM. Quantitative magnetic resonance first-pass perfusion analysis: inter- and intraobserver agreement. J Cardiovasc Magn Reson. 2001;3(3):247-56. doi: 10.1081/jcmr-100107473. PMID 11816621